CLINICAL TRIAL: NCT03691246
Title: Research on Burden of Disease for Patients With Myocardial Infarction Combining Dyslipidemia in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Cardiovascular Association (Other)
Collaborators: Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Shanghai Zhongshan Hospital (Other); Guangdong Provincial People's Hospital (Other); Sichuan Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GUSU17003
Record Dates: First submitted 2018-09-22; First posted 2018-10-01 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-11

CONDITIONS: Myocardial Infarction; Dyslipidemias
Keywords: Myocardial Infarction; Dyslipidemia
MeSH Terms: conditions — Myocardial Infarction; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is medical record review and questionnaire survey on the economic burden on Chinese patients with myocardial infarction accompanied by dyslipidemia in a real-world environment.

The primary objective of the study is to investigate the economic burden of disease on patients and the factors influencing it, which may include the mode of treatment for dyslipidemia, drugs for the secondary prevention of myocardial infarction, the outcome of treatment for dyslipidemia, adverse drug reactions and major cardiovascular events.

The secondary objectives of the study include:

1. patient compliance with medication;
2. health-related quality of life (HRQoL) in patients.

DETAILED DESCRIPTION:
This study is a multicenter retrospective cohort survey study using a cross-sectional design. It is conducted mainly by a medical record review, questionnaire survey and medical examination to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Patients were hospitalized because of acute myocardial infarction in a study hospital between January 1, 2016 and December 31, 2016. If a patient was hospitalized because of multiple occurrences of myocardial infarction during this period, his/her initial hospitalization because of myocardial infarction will be considered index hospitalization. Patients undergo continuous screening in a reverse order based on time.
* Patients did not die during "index hospitalization".
* Patients had Low-density lipoprotein≥1.8 mmol/L shown by the first measurement of blood lipids or were using lipid-regulating drugs at the first measurement of blood lipids during "index hospitalization" in 2016.
* Patients consent to participate in this study and grant informed consent; or the family of a patient who died before telephone screening consents to provide relevant information and grant informed consent.

Exclusion Criteria:

* Patients participated in interventional clinical trials after "index hospitalization".
* Patients had paid <5 visits to the outpatient clinics of a study hospital within one year since discharge after "index hospitalization" (if patients who have died within one year since discharge after "index hospitalization").
* There is a barrier to communication with a patient or his/her family (if the patient has died); a patient or his/her family (if the patient has died) cannot correctly understand and answer questions normally.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were hospitalized because of acute myocardial infarction in a study hospital between January 1, 2016 and December 31, 2016. If a patient was hospitalized because of multiple occurrences of myocardial infarction during this period, his/her initial hospitalization because of myocardial infarction will be considered index hospitalization. Patients undergo continuous screening in a reverse order based on time.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Economic burden of disease | 2 to 3 years
  Total of costs for outpatient/emergency visits after discharge since "index hospitalization" (e.g., registration fees, examination fees, inspection fees, charges for drugs and other expenses), inpatient expenses (e.g., charges for percutaneous coronary intervention /coronary artery bypass graft, bed fees, charges for drugs, charges for materials, charges for nursing care and other expenses), payments for health care workers, fees for transportation, fees for accommodation and food, costs due to losses of time and capacity for physical labor for patients and their families, charges for visits to other medical institutions due to dyslipidemia and related diseases, as well as expenses for medications and health products purchased from drug stores.

SECONDARY OUTCOMES:
Health-related quality of life | 2 to 3 years
  The EuroQol five dimensions questionnaire with three-level (EQ-5D-3L) scores are calculated using the scoring system for the Chinese population. Then, the mean and standard deviation of health utility values (HUVs) are reported.
  EQ-5D-3L is a standardized instrument for use as a measure of health outcome. The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1 point), some problems (2 points), extreme problems (3 points).
patient compliance with medication | 2 to 3 years
  Medication compliance is reported mainly based on the frequency of oral administration on time and the percentage of patients taking drugs on time, which are assessed by patients themselves in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, master, Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Bays HE, Chapman RH, Fox KM, Grandy S; SHIELD Study Group. Comparison of self-reported survey (SHIELD) versus NHANES data in estimating prevalence of dyslipidemia. Curr Med Res Opin. 2008 Apr;24(4):1179-86. doi: 10.1185/030079908x280527. Epub 2008 Mar 14. PMID 18346311
- [Background] Joffres M, Shields M, Tremblay MS, Connor Gorber S. Dyslipidemia prevalence, treatment, control, and awareness in the Canadian Health Measures Survey. Can J Public Health. 2013 Apr 24;104(3):e252-7. doi: 10.17269/cjph.104.3783. PMID 23823891
- [Background] Alhabib KF, Sulaiman K, Al-Motarreb A, Almahmeed W, Asaad N, Amin H, Hersi A, Al-Saif S, AlNemer K, Al-Lawati J, Al-Sagheer NQ, AlBustani N, Al Suwaidi J; Gulf RACE-2 investigators. Baseline characteristics, management practices, and long-term outcomes of Middle Eastern patients in the Second Gulf Registry of Acute Coronary Events (Gulf RACE-2). Ann Saudi Med. 2012 Jan-Feb;32(1):9-18. doi: 10.5144/0256-4947.2012.9. PMID 22156634
- [Background] Tuppin P, Riviere S, Rigault A, Tala S, Drouin J, Pestel L, Denis P, Gastaldi-Menager C, Gissot C, Juilliere Y, Fagot-Campagna A. Prevalence and economic burden of cardiovascular diseases in France in 2013 according to the national health insurance scheme database. Arch Cardiovasc Dis. 2016 Jun-Jul;109(6-7):399-411. doi: 10.1016/j.acvd.2016.01.011. Epub 2016 Apr 11. PMID 27079468
- [Background] Mota D, Mattos AC, Oliveira G, Avezum A. The Need for Brazil to Focus on CVD. Glob Heart. 2016 Dec;11(4):439-440. doi: 10.1016/j.gheart.2016.10.001. No abstract available. PMID 27938835
- [Background] Moran A, Gu D, Zhao D, Coxson P, Wang YC, Chen CS, Liu J, Cheng J, Bibbins-Domingo K, Shen YM, He J, Goldman L. Future cardiovascular disease in china: markov model and risk factor scenario projections from the coronary heart disease policy model-china. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):243-52. doi: 10.1161/CIRCOUTCOMES.109.910711. Epub 2010 May 4. PMID 20442213
- [Background] Authors/Task Force Members:; Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WM, Vlachopoulos C, Wood DA, Zamorano JL. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias: The Task Force for the Management of Dyslipidaemias of the European Society of Cardiology (ESC) and European Atherosclerosis Society (EAS) Developed with the special contribution of the European Assocciation for Cardiovascular Prevention & Rehabilitation (EACPR). Atherosclerosis. 2016 Oct;253:281-344. doi: 10.1016/j.atherosclerosis.2016.08.018. Epub 2016 Sep 1. No abstract available. PMID 27594540